CLINICAL TRIAL: NCT03984136
Title: The Effectiveness of HIV Results Exchange Mechanism on Promoting Testing Behavior Among Men Who Have Sex With Men: A Cluster Randomized Controlled Trial
Brief Title: HIV Results Exchange Mechanism on Promoting HIV Testing Among MSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Chun Hao, Associate Professor of School of Public Health, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: No.054 of ethic committee
Record Dates: First submitted 2019-06-09; First posted 2019-06-12 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: HIV/AIDS
Keywords: HIV testing; Men who have sex with men
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Men will be required to exchange the Center for Disease Control and Prevention certified online HIV results (COHIV) with friends conditionally.
  Interventions: Behavioral: COHIV with exchange mechanism
- Control group (Active Comparator): Men will share the Center for Disease Control and Prevention certified online HIV results (COHIV) with friends freely without conditional exchange requirement.
  Interventions: Behavioral: COHIV without exchange mechanism

INTERVENTIONS:
Behavioral: COHIV with exchange mechanism — A WeChat-based mini program has been developed to send and receive Center for Disease Control and Prevention certified online HIV results (COHIV). WeChat is the ubiquitous communication and social networking tool in China. Participants in the intervention group will receive his friend's COHIV only when the participants share their own in exchange. If the participant already has the COHIV, the system will lead the user to send his COHIV to the friend. If the participant does not have the COHIV, the system will guide him to make online appointment at the testing clinic.
  Arms: Intervention group
Behavioral: COHIV without exchange mechanism — The participants in the control group will be able to receive the friend's Center for Disease Control and Prevention certified online HIV results (COHIV) entirely at the friend's discretion without the mandatory exchange requirement. The system will also guide users on how to get an HIV test by making appointments with the MSM friendly clinics in the mini program.
  Arms: Control group

SUMMARY:
This will be a two-arm cluster randomized controlled trial. The control group can share their Center for Disease Control and Prevention certified online HIV results (COHIV) with another party freely through a social networking tool, while the intervention group will be asked for the COHIV before he can see the COHIV of his friend. The investigators hypothesize that the requires exchange will promote HIV testing and thus reduce HIV incidence among MSM.

DETAILED DESCRIPTION:
This will be a two-arm cluster randomized controlled trial. A WeChat-based mini program has been developed to send and receive Center for Disease Control and Prevention certified online HIV results (COHIV). WeChat is the ubiquitous communication and social networking tool in China. We will use the social network method for participant recruitment. A social network consists of one ego and some alters, and in this study a social network will be considered as a cluster. In a social network, ego is the MSM who shares his certified HIV test results with or without exchange mechanism by the WeChat mini program, while alters are recipients of the shared links. So the ego can shares his COHIV with many alters. After an ego shares the certified HIV test result with exchange mechanism (intervention group) or without exchange mechanism (control group) with their WeChat contactors, the people who click the link will be candidate alters in our study. 1020 alters will be recruited as the participants and the randomization would be based on the unit of social network, which means the alters will be randomized into the same group that the ego is in.

Participants in the intervention group will receive his friend's COHIV and can only open it when the participants share their own in exchange. If the participant already has the COHIV, the system will lead the user to send his COHIV to the friend. If the participant does not have the COHIV, the system will guide him to make online appointment at the testing clinic. The participants in the control group will be able to receive and open the friend's COHIV entirely at the friend's discretion without the mandatory exchange requirement. The system will also guide users on how to get an HIV test by making appointments with the MSM friendly clinics in the mini program. Questionnaires are scheduled at baseline, month 3, 6 and 9. Follow-up questionnaires will be delivered through WeChat. The primary outcome is HIV testing rate of the participants in the past three months.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than18 years old
* Had anal sex with men
* HIV unknown or negative
* Plan to live in Guangzhou for the next year

Exclusion Criteria:

- Cannot complete questionnaire survey due to difficulty in reading or communication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1008 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with self-reported HIV testing in the past three months | Enrollment time
  Self-reported HIV testing includes any classification of HIV testing, will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV testing in the past three months | 3 months after enrollment
  Self-reported HIV testing includes any classification of HIV testing, will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV testing in the past three months | 6 months after enrollment
  Self-reported HIV testing includes any classification of HIV testing, will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV testing in the past three months | 9 months after enrollment
  Self-reported HIV testing includes any classification of HIV testing, will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV self-testing(HIVST) in the past three months | Enrollment time
  HIVST will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV self-testing(HIVST) in the past three months | 3 months after enrollment
  HIVST will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV self-testing(HIVST) in the past three months | 6 months after enrollment
  HIVST will be measured by self-reported data from online questionnaires.
Number of participants with self-reported HIV self-testing(HIVST) in the past three months | 9 months after enrollment
  HIVST will be measured by self-reported data from online questionnaires.
Number of participants with clinic-based HIV testing services (HTS) in the past three months | Enrollment time
  Clinic-based HTS will be measured by the objectively recorded HIV testing at the HIV clinic which will be captured real-time through the computer system.
Number of participants with clinic-based HIV testing services (HTS) in the past three months | 3 months after enrollment
  Clinic-based HTS will be measured by the objectively recorded HIV testing at the HIV clinic which will be captured real-time through the computer system.
Number of participants with clinic-based HIV testing services (HTS) in the past three months | 6 months after enrollment
  Clinic-based HTS will be measured by the objectively recorded HIV testing at the HIV clinic which will be captured real-time through the computer system.
Number of participants with clinic-based HIV testing services (HTS) in the past three months | 9 months after enrollment
  Clinic-based HTS will be measured by the objectively recorded HIV testing at the HIV clinic which will be captured real-time through the computer system.

SECONDARY OUTCOMES:
Number of participants with sexually transmitted diseases (STDs) testing | Enrollment time
  Sexually transmitted diseases (STDs) testing will be measured by self-reported data from online questionnaires and registered data in the HIV testing system.
Number of participants with sexually transmitted diseases (STDs) testing | 3 months after enrollment
  Sexually transmitted diseases (STDs) testing will be measured by self-reported data from online questionnaires and registered data in the HIV testing system.
Number of participants with sexually transmitted diseases (STDs) testing | 6 months after enrollment
  Sexually transmitted diseases (STDs) testing will be measured by self-reported data from online questionnaires and registered data in the HIV testing system.
Number of participants with sexually transmitted diseases (STDs) testing | 9 months after enrollment
  Sexually transmitted diseases (STDs) testing will be measured by self-reported data from online questionnaires and registered data in the HIV testing system.
Sexual behaviors in the past three months | Enrollment time
  High-risk and protective sexual behaviors include regular or casual sex partners; request for disclosure of HIV status before sex in the past 3 months; unprotected anal intercourse (UAI) with sex partners in the past 3 months; HIV testing service appointment and HIV test results, will be measured by self-reported data from online questionnaires and the routinely collect data in the HIV testing service system.
Sexual behaviors in the past three months | 3 months after enrollment
  High-risk and protective sexual behaviors include regular or casual sex partners; request for disclosure of HIV status before sex in the past 3 months; unprotected anal intercourse (UAI) with sex partners in the past 3 months; HIV testing service appointment and HIV test results, will be measured by self-reported data from online questionnaires and the routinely collect data in the HIV testing service system.
Sexual behaviors in the past three months | 6 months after enrollment
  High-risk and protective sexual behaviors include regular or casual sex partners; request for disclosure of HIV status before sex in the past 3 months; unprotected anal intercourse (UAI) with sex partners in the past 3 months; HIV testing service appointment and HIV test results, will be measured by self-reported data from online questionnaires and the routinely collect data in the HIV testing service system.
Sexual behaviors in the past three months | 9 months after enrollment
  High-risk and protective sexual behaviors include regular or casual sex partners; request for disclosure of HIV status before sex in the past 3 months; unprotected anal intercourse (UAI) with sex partners in the past 3 months; HIV testing service appointment and HIV test results, will be measured by self-reported data from online questionnaires and the routinely collect data in the HIV testing service system.
HIV testing norms | Enrollment time
  HIV testing norms are measured using six survey items that are each on a four-point Likert scale in online surveys. All six items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate less positive HIV testing social norms.
HIV testing norms | 3 months after enrollment
  HIV testing norms are measured using six survey items that are each on a four-point Likert scale in online surveys. All six items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate less positive HIV testing social norms.
HIV testing norms | 6 months after enrollment
  HIV testing norms are measured using six survey items that are each on a four-point Likert scale in online surveys. All six items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate less positive HIV testing social norms.
HIV testing norms | 9 months after enrollment
  HIV testing norms are measured using six survey items that are each on a four-point Likert scale in online surveys. All six items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate less positive HIV testing social norms.
HIV stigma | Enrollment time
  HIV stigma will be measured by a 7-item version of the HIV stigma scale, designed to measure the extent to which participants anticipated negative interpersonal and interpersonal consequences were they to contract HIV in the future. All seven items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate greater stigma.
HIV stigma | 3 months after enrollment
  HIV stigma will be measured by a 7-item version of the HIV stigma scale, designed to measure the extent to which participants anticipated negative interpersonal and interpersonal consequences were they to contract HIV in the future. All seven items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate greater stigma.
HIV stigma | 6 months after enrollment
  HIV stigma will be measured by a 7-item version of the HIV stigma scale, designed to measure the extent to which participants anticipated negative interpersonal and interpersonal consequences were they to contract HIV in the future. All seven items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate greater stigma.
HIV stigma | 9 months after enrollment
  HIV stigma will be measured by a 7-item version of the HIV stigma scale, designed to measure the extent to which participants anticipated negative interpersonal and interpersonal consequences were they to contract HIV in the future. All seven items were rated on a Likert-type scale (1=Strongly Disagree; 4=Strongly Agree). The mean score is reported, ranged from 1 to 4. Higher values indicate greater stigma.
Risk perception of HIV in MSM community | Enrollment time
  Risk perception of HIV in MSM community will be measured by self-perceived HIV prevalence in the circle.
Risk perception of HIV in MSM community | 3 months after enrollment
  Risk perception of HIV in MSM community will be measured by self-perceived HIV prevalence in the circle.
Risk perception of HIV in MSM community | 6 months after enrollment
  Risk perception of HIV in MSM community will be measured by self-perceived HIV prevalence in the circle.
Risk perception of HIV in MSM community | 9 months after enrollment
  Risk perception of HIV in MSM community will be measured by self-perceived HIV prevalence in the circle.
HIV report delivery | Enrollment time
  HIV report delivery includes the proportion of Egos who forward and read their reports; the proportion of Alters who receive and read egos' reports; the proportion of alters who get their own HIV reports; the proportion of forwarded report usage among MSM and the satisfaction of online HIV report service. These data will be collected by the WeChat-based data portal.
HIV report delivery | 3 months after enrollment
  HIV report delivery includes the proportion of Egos who forward and read their reports; the proportion of Alters who receive and read egos' reports; the proportion of alters who get their own HIV reports; the proportion of forwarded report usage among MSM and the satisfaction of online HIV report service. These data will be collected by the WeChat-based data portal.
HIV report delivery | 6 months after enrollment
  HIV report delivery includes the proportion of Egos who forward and read their reports; the proportion of Alters who receive and read egos' reports; the proportion of alters who get their own HIV reports; the proportion of forwarded report usage among MSM and the satisfaction of online HIV report service. These data will be collected by the WeChat-based data portal.
HIV report delivery | 9 months after enrollment
  HIV report delivery includes the proportion of Egos who forward and read their reports; the proportion of Alters who receive and read egos' reports; the proportion of alters who get their own HIV reports; the proportion of forwarded report usage among MSM and the satisfaction of online HIV report service. These data will be collected by the WeChat-based data portal.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Hao, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Lingnan Partner Community Support Centre, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data that underlie the results in the published article would be available from the principal investigator on reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Sun HT, Fan XR, Gu YZ, Lu YH, Qiu JL, Yang QL, Li JH, Gu J, Hao C. WeChat-Based HIV e-Report, a New Approach for HIV Serostatus Requests and Disclosures Among Men Who Have Sex With Men: Prospective Subgroup Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 May 8;11:e44513. doi: 10.2196/44513. PMID 37155223
- [Derived] Shi Y, Qiu J, Yang Q, Chen T, Lu Y, Chen S, Fan X, Lin Z, Han Z, Lu J, Qian H, Gu J, Xu DR, Gu Y, Hao C. Increasing the HIV testing among MSM through HIV test result exchange mechanism: study protocol for a cluster randomized controlled trial. BMC Infect Dis. 2021 Aug 6;21(1):764. doi: 10.1186/s12879-021-06484-y. PMID 34362323